CLINICAL TRIAL: NCT00224185
Title: Evaluation of the Lungs of Normal Individuals With Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing and Bronchial Wall Biopsy
Brief Title: Evaluation of Lungs of Normal Individuals by Lung Lavage, Brushing and Bronchial Wall Biopsy
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York Presbyterian Hospital (Other); Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB0005004439; NCT00234325 (obsolete NCT alias)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Smoking; Lung Diseases
Keywords: Healthy individuals; smokers; ex-smokers; non-smokers
MeSH Terms: conditions — Smoking; Lung Diseases; Smoking Cessation | interventions — Bronchoalveolar Lavage; Bronchoalveolar Lavage Fluid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens will be retained from both a blood draw and a bronchial wall biopsy which obtains tissue to a depth of 2-3 mm and includes epithelial and subepithelial tissue.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Bronchopulmonary Lung Lavage — Lung Lavage is a Washing. Bronchoscopy consists of the passage via the mouth or nose of a flexible fiberoptic bronchoscopy into the airways. During the lavage (washing) procedure, sterile 0.9% saline (5 x 20 ml aliquots in 1 to 3 sites) is instilled into the lung and immediately suctioned back, washing off cells lining the airways. Once the fluid has been collected, the fluid is centrifuged and the cells are collected and counted.
  Other Names: Bronchoalveolar Lavage
Procedure: Bronchial Brushing — Bronchoscopy consists of the passage via the mouth or nose of a flexible fiberoptic bronchoscopy into the airways. During the brushing procedure, a small cytology brush is passed through the bronchoscope, and a small area of the airway wall is brushed gently (in up to 20 different sites in the large and small airways) to obtain epithelial cells lining the airway. Cells collected by airway brushing will be washed, counted, and evaluated for viability. They will also be studied for differential cell count by standard procedures. Collected airway cells will be used to carry out studies assess expression of various genes and to study viral gene transfer.
  Other Names: Bronchial Washing
Procedure: Bronchial Wall Biopsy — This is a safe and widely used investigative method in pulmonary medicine. In this procedure, a small biopsy forceps is passed through the bronchoscope and, under direct vision, a small biopsy (in up to 5 sites) is obtained from the bronchial wall. A biopsy obtains tissue to a depth of 2-3 mm, and includes epithelial and subepithelial tissue.
  Other Names: Lung Biopsy

SUMMARY:
The purpose of this study is to obtain biologic materials from the blood and lungs of normal individuals to establish a set of normal range for various parameters. These will provide important information when applied to individuals with various pulmonary diseases, and will help in understanding of the etiology and pathogenesis of various lung diseases.

DETAILED DESCRIPTION:
Study procedures will be performed at the Weill Cornell Medical College-New York Presbyterian Hospital and/or Weill Greenburg York Avenue Building. Study procedures done elsewhere that are within the protocol timeframe will be accepted if seen fit by the investigators so that they are not repeated unnecessarily. Study individuals who undergo bronchoscopy with intravenous administration of sedatives and analgesia may be required to stay overnight. Bronchoscopy is normally an ambulatory procedure. The subject is observed after the bronchoscopy, including vital signs and level of consciousness, until they are back to baseline. An overnight stay would only be required if the individual was not, in the judgment of the attending physician, safe to be discharged as is standard practice. Follow up of all participants are carried out by telephone within 1 wk following the procedure.

Rockefeller University has been added as a second site.

Individuals undergoing bronchoscopy without intravenous administration of sedatives and analgesia are not required to stay overnight due to the lack of administration of CNS-altering drugs and the limited sampling involved (tracheal brushes only).

ELIGIBILITY:
Inclusion Criteria:

* All study subjects should be able to provide informed consent
* Males or females ages 18 years and older.
* Must provide HIV informed consent.
* Non-smokers, ex-smokers and smokers.

Exclusion Criteria:

* Individuals not deemed in good overall health by the investigator will not be accepted into the study.
* Drug and/or alcohol abuse within the past six months.
* Individuals with history of chronic lung disease, including asthma or with recurrent or recent (within three months) acute pulmonary disease will not be accepted into the study.
* Individuals with allergies to atropine or any local anesthetic will not be accepted into the study.
* Individuals with allergies to pilocarpine, isoproterenol, terbutaline, atropine or aminophylline will not be accepted into the study
* Females who are pregnant or nursing will not be accepted into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The source of potential subjects will be the population of 'normal', as defined by the eligibility criteria below, individuals in the New York metropolitan area and elsewhere. Up to one hundred volunteers will take part in the study each year. Accrual will be random with no bias as to gender or racial/ethnic group. All study individuals will be males or females that are 18 years or older and are able to provide informed consent. Advertisements will be posted at various educational institutions and hospitals and placed in newspapers in the New York metropolitan area. Paid volunteer referrals will also be used for patient recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2004-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Evaluate etiology of lung diseases | 9/31/2012
  We hope to learn more about the specific causes of lung disease, how lung disease manifests and progresses, and how lung disease can be treated.

SECONDARY OUTCOMES:
Effect of smoking on the genes of airway epithelial cells | 9/31/2012
  We hope to learn how smoking affects the genetic composition of the cells that line the airways (windpipes) of the lungs, and whether there are differences in the genetic composition of the cells that line the windpipe in normal individuals who smoke.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Department of Genetic Medicine, Weill Cornell Medical College
Locations (1):
- Department of Genetic Medicine, WMC of Cornell Univeristy, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang G, Wang R, Ferris B, Salit J, Strulovici-Barel Y, Hackett NR, Crystal RG. Smoking-mediated up-regulation of GAD67 expression in the human airway epithelium. Respir Res. 2010 Oct 29;11(1):150. doi: 10.1186/1465-9921-11-150. PMID 21034448
- [Derived] Carolan BJ, Harvey BG, Hackett NR, O'Connor TP, Cassano PA, Crystal RG. Disparate oxidant gene expression of airway epithelium compared to alveolar macrophages in smokers. Respir Res. 2009 Nov 17;10(1):111. doi: 10.1186/1465-9921-10-111. PMID 19919714